CLINICAL TRIAL: NCT05894577
Title: ACTIV-6: COVID-19 Outpatient Randomized Trial to Evaluate Efficacy of Repurposed Medications
Brief Title: ACTIV-6: COVID-19 Study of Repurposed Medications - Arm F (Montelukast)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Susanna Naggie, MD (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Susanna Naggie, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00107921_F; 3U24TR001608-05W1 (NIH)
Record Dates: First submitted 2023-06-06; First posted 2023-06-08 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Covid19
Keywords: SARS-CoV-2; COVID-19; Placebo; Duke University Health System; Outcomes; Duke Clinical Research Institute; ACTIV 6; ACTIV; montelukast
MeSH Terms: conditions — COVID-19 | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: Double-Blind, Placebo-Controlled, Randomized Trial
Who Masked: Participant, Care Provider
Masking Description: The participant and study teams will know which study drug the participant is allocated to, but will be blinded to study drug versus placebo because they will be matching.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm F - Montelukast (Experimental): Montelukast will be self-administered orally by each participant at a dose of 10 mg once a day for 14 days.
  Interventions: Drug: Montelukast
- Arm F - Placebo (Placebo Comparator): Placebo - appearance and size matched to active study drug.
  Placebo will be self-administered orally by each participant, with number of tablets matched to active study drug dosing.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Each study arm will contain a placebo comparator. Placebo will look similar to study drug and will be administered via the same route of administration and dose. However, placebo will be an inactive substance, containing no study drug.
  Arms: Arm F - Placebo
Drug: Montelukast — Montelukast sodium is a white to off-white powder. The 10 mg montelukast tablets are beige, rounded square-shaped, biconvex, film-coated tablets. Each tablet contains 10.4 mg of montelukast sodium, which is equivalent to 10 mg montelukast. All packaging will be labeled to indicate that the product is for investigational use.
  Arms: Arm F - Montelukast

SUMMARY:
The purpose of this study is to evaluate the effectiveness of repurposed medications (study drug(s) in reducing symptoms of non-hospitalized participants with mild to moderate COVID-19. Participants will receive either study drug or placebo. They will self-report any new or worsening symptoms or medical events they may experience while taking study drug or placebo. This study is intended to be all remote with no in person visits, unless the study team feels it is in the best interest of a participant to see them in person.

Prior and current drug arms are listed on clinicaltrials.gov and will be updated with the activation of any new drug arms. Each study arm will also have its own clinicaltrials.gov entry and will include "Pro00107921" in the Unique Protocol ID.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a novel betacoronavirus that first emerged in December 2019 and has since caused a global pandemic unseen in almost a century with respect to the number of cases and overall mortality. The clinical disease related to SARS-CoV-2 is referred to as Coronavirus Disease 2019 (COVID-19). Over 2020, advances were made for treatment of COVID-19 and several vaccinations have received emergency use authorization for prevention of SARS-CoV-2 infections. However, the pandemic continues to evolve with new variants and surges of infections in different regions of the world, requiring an ongoing evidence-generating platform, in particular for the treatment of COVID-19 infection in the outpatient setting.

This proposed platform protocol can serve as an evidence generating system for prioritized drugs repurposed from other indications with an established safety record and preliminary evidence of clinical efficacy for the treatment of COVID-19. The ultimate goal is to evaluate if repurposed medications can make participants feel better faster and reduce death and hospitalization.

This platform protocol is designed to be flexible so that it is suitable for a wide range of settings within healthcare systems and in community settings where it can be integrated into routine COVID-19 testing programs and subsequent treatment plans. This platform protocol will enroll participants in an outpatient setting with a confirmed polymerase chain reaction (PCR) or antigen test for SARS-CoV-2.

Participants will be randomized to study drugs or placebo based on the arms that are actively enrolling at the time of randomization. Study drugs may be added or removed according to adaptive design and/or emerging evidence. When there are multiple study drugs available, randomization will occur based on appropriateness of each drug for the participant as determined by the study protocol and investigator and participant equipoise. Each participant will be required to randomize to at least one study drug versus placebo. The probability of placebo to treatment will remain the same regardless of eligibility decisions.

Eligible participants will be randomized (1:1), in a blinded fashion, to either the study drug arm or placebo arm in addition to standard of care. As additional study drugs are added, the randomization will be altered to leverage placebo data across arms. Participants will receive a complete supply study drug or placebo with the quantity depending on the study drug/placebo to which they are randomized.

All study visits are designed to be remote. However, screening and enrollment may occur in-person at sites and unplanned study visits may occur in-person or remotely, as deemed appropriate by the site investigator for safety purposes. Participants will be asked to complete questionnaires and report safety events during the study. Participants will be prompted by the online system to report safety events and these will be reviewed and confirmed via medical records and site staff, as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Completed Informed Consent
* Age ≥ 30 years old
* Confirmed SARS-CoV-2 infection (or reinfection) by any authorized or approved polymerase chain reaction (PCR) or antigen test collected within 10 days of screening
* Two or more current symptoms of acute infection for ≤7 days. Symptoms include the following: fatigue, dyspnea, fever, cough, nausea, vomiting, diarrhea, body aches, chills, headache, sore throat, nasal symptoms, new loss of sense of taste or smell

Exclusion Criteria:

* Prior diagnosis of COVID-19 infection (> 10 days from screening)
* Current or recent (within 10 days of screening) hospitalization
* Known allergy/sensitivity or any hypersensitivity to components of the study drug or placebo
* Known contraindication(s) to study drug including prohibited concomitant medications

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1453 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Naggie, MD, Principal Investigator — Duke Clinical Research Institute; Adrian Hernandez, MD, Principal Investigator — Duke Clinical Research Institute
Locations (109):
- United States (109):
  - Chandler Regional Medical Center, Chandler, Arizona
  - Lamb Health, LLC, Gilbert, Arizona
  - First Care Medical Clinic, Mesa, Arizona
  - Trident Health Center, Peoria, Arizona
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Assuta Family Medical Group APMC, North Hollywood, California
  - Stanford, Palo Alto, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Doctors Medical Group of Colorado Springs, P.C., Colorado Springs, Colorado
  - Pine Ridge Family Medicine Inc., Colorado Springs, Colorado
  - Tabitha B. Fortt, M.D., LLC, Stamford, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Arena Medical Group, Deerfield Beach, Florida
  - Lupus Foundation of Gainesville, Gainesville, Florida
  - University of Florida Health, Gainesville, Florida
  - L and A Morales Healthcare, Inc, Hialeah, Florida
  - University of Florida-JAX-ASCENT, Jacksonville, Florida
  - AMRON Vitality and Wellness Center, LLC, Jacksonville, Florida
  - Sunshine Walk In Clinic, Lake Mary, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - The Angel Medical Research Corporation, Miami Lakes, Florida
  - Innovation Clinical Trials Inc., Palmetto Bay, Florida
  - Lice Source Services Plantation, Plantation, Florida
  - Premier Health, St. Petersburg, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - UF Health Precision Health Research, The Villages, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory Healthcare, Atlanta, Georgia
  - Essential Medical Care, Inc., College Park, Georgia
  - Clincept, LLC, Columbus, Georgia
  - HOPE Clinical Research and Wellness, Conyers, Georgia
  - David Kavtaradze MD, Inc., Cordele, Georgia
  - Elite Family Practice, Douglasville, Georgia
  - Christ the King Health Care, P.C., Loganville, Georgia
  - Miller Family Practice, LLC, Macon, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Olivo Wellness Medical Center, Chicago, Illinois
  - NorthShore Medical Group, Evanston, Illinois
  - Advanced Medical Care, Ltd, Lake Zurich, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Franciscan Health Michigan City, Michigan City, Indiana
  - Del Pilar Medical and Urgent Care, Mishawaka, Indiana
  - University of Kansas - Wichita, Wichita, Kansas
  - A New Start II, LLC, Central City, Kentucky
  - Christus Saint Frances Hospita, Alexandria, Louisiana
  - University Medical Center- New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Jadestone Clinical Research, LLC, Rockville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Health Quality Primary Care, Lawrence, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Ananda Medical Clinic, Dearborn, Michigan
  - GFC of Southeastern Michigan, PC, Detroit, Michigan
  - Romancare Health Services, Detroit, Michigan
  - Essentia Health, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri - Columbia, Columbia, Missouri
  - Comprehensive Pain Management and Endocrinology, Henderson, Nevada
  - Focus Clinical Research Solutions, Bayonne, New Jersey
  - Raritan Bay Primary Care & Cardiology Associates, Matawan, New Jersey
  - G&S Medical Associates, LLC, Paterson, New Jersey
  - Mediversity Healthcare, Turnersville, New Jersey
  - Christus St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - Geriatrics and Medical Associates, Clinton, New York
  - Weill Cornell Medical College, New York, New York
  - Spinal Pain and Medical Rehab, PC, Yonkers, New York
  - Vaidya MD PLLC, Clayton, North Carolina
  - Maria Medical Center, PLLC, Dunn, North Carolina
  - Duke Clinical Research Institute, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Lapis Clinical Research, Mooresville, North Carolina
  - Superior Clinical Research, Smithfield, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Diabetes and Endocrinology Assoc. of Stark County, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - TriHealth, Inc, Montgomery, Ohio
  - The Heart and Medical Center, Durant, Oklahoma
  - Hugo Medical clinic, Hugo, Oklahoma
  - Ascension St. John, Tulsa, Oklahoma
  - Bucks County Clinical Research, Morrisville, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical Trials Center of Middle TN, Franklin, Tennessee
  - Rapha Family Wellness, Hendersonville, Tennessee
  - Medical Specialists of Knoxville, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Express Family Clinic, Allen, Texas
  - DHR Health Institute for Research, Edinburg, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - Highlands Medical Associates, P.A., Highlands, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Family Practice Doctors P.A., Humble, Texas
  - Texas Health Physicians Group, Irving, Texas
  - Kintex Group Texas LLC, DBA Activian Clinical Research, Kingwood, Texas
  - University Diagnostics and Treatment Clinic, Pasadena, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Jeremy W. Szeto, D.O., P.A., Sugar Land, Texas
  - University of Texas Rio Grande Valley, Weslaco, Texas
  - University of Virginia, Charlottesville, Virginia
  - Providence Medical Research Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will share this data after it has been de-identified. We will share data beginning around 6 months after publication and for up to 36 months afterward. Access will only be shared with those who have obtained prior IRB approval to be able to access this data.
Supporting Information: SAP, CSR
Time Frame: Up to 36 months after publication
Access Criteria: Interested investigators will need to seek prior IRB approval before access to any data is granted.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm F - Placebo: Placebo - appearance and size matched to active study drug.
  Placebo will be self-administered orally by each participant, with number of tablets matched to active study drug dosing.
  Placebo: Each study arm will contain a placebo comparator. Placebo will look similar to study drug and will be administered via the same route of administration and dose. However, placebo will be an inactive substance, containing no study drug.
Period: Overall Study
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Started | 741 | 712
Completed | 628 | 622
Not Completed | 113 | 90
Not completed — No receipt of study drug | 14 | 13
Not completed — Randomized not enrolled (Drug not received) | 11 | 14
Not completed — Screen Fail | 2 | 0
Not completed — Study drug recall | 86 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm F - Montelukast | Arm F - Placebo | Total
Number analyzed (Participants) | 628 | 622 | 1250
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [42 to 61] | 54 [43 to 62] | 53 [42 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 388 | 365 | 753
  Male | 240 | 257 | 497
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 415 | 392 | 807
  Not Hispanic or Latino | 213 | 230 | 443
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 1 | 3
  Race: Asian | 20 | 22 | 42
  Race: Black, African American, or African | 84 | 70 | 154
  Race: Middle Eastern or North African | 8 | 10 | 18
  Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Race: White | 483 | 484 | 967
  Race: More than one race | 5 | 7 | 12
  Race: None of the above | 16 | 19 | 35
  Race: Prefer not to answer | 7 | 6 | 13
  Race: No response | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 628 | 622 | 1250

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Recovery in Days
Description: Time to sustained recovery was the number of days between receipt of study drug and the third of 3 consecutive days without symptoms. Participants who died, by definition, did not recover regardless of reported symptom freedom. The reported summary is the median survival time.
Time Frame: Up to 28 days
Population: Participants with data collected.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 619 | 613
days | 10 [10 to 11] | 10 [10 to 11]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Test type: Superiority — Posterior probability of efficacy (P(HR>1)); Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.92 to 1.12] — The interval is a highest-density credible interval. Adjustment variables: randomization, age, sex, duration of symptoms prior to study drug, calendar time, vaccination status, geographic region, call center indicator, and baseline symptom severity

2. Secondary Outcome: Number of Participants With Hospitalization or Death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
Participants | 2 | 2
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; No hypothesis test or decision rule was evaluated; Test type: Superiority; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.14 to 7.07] — Low event rate precluded covariate adjustment

3. Secondary Outcome: Number of Participants With Mortality
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
Participants | 0 | 0

4. Secondary Outcome: Time to Mortality
Description: Time to mortality was the number of days between drug receipt and death.
Time Frame: Up to 28 days
Population: Data not collected as no participants experienced mortality.
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Hospitalization, Urgent Care, Emergency Room Visit, or Death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
Participants | 18 | 18
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; No hypothesis test or decision rule was evaluated; Test type: Superiority — Posterior probability of efficacy (P(HR<1)); Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.45 to 1.84] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants at Each Score on the COVID Clinical Progression Scale at Day 7
Description: COVID Clinical Progression Scale is a scale of 0 to 8 where 0 = No clinical or virological evidence of infection, 1 = No limitation of activities, 2 = Limitation of activities, 3 = Hospitalized, no oxygen therapy, 4 = Hospitalized, on oxygen by mask or nasal prongs, 5 = Hospitalized, on non-invasive ventilation or high-flow oxygen, 6 = Hospitalized, on intubation and mechanical ventilation, 7 = Hospitalized, on ventilation + additional organ support (pressors, RRT, ECMO), 8 = Death.
Time Frame: Day 7
Population: Participants with data collected at day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 606 | 602
Participants
  0 = No clinical or virological evidence of infection | 22 | 28
  1 = No limitation of activities | 564 | 557
  2 = Limitation of activities | 20 | 17
  3 = Hospitalized, no oxygen therapy | 0 | 0
  4 = Hospitalized, on oxygen by mask or nasal prongs | 0 | 0
  5 = Hospitalized, on non-invasive ventilation or high-flow oxygen | 0 | 0
  6 = Hospitalized, on intubation and mechanical ventilation | 0 | 0
  7 = Hospitalized, on ventilation + additional organ support | 0 | 0
  8 = Death | 0 | 0
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; No hypothesis test or decision rule was evaluated; Test type: Superiority — Posterior probability of efficacy (P(OR<1)); Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.50 to 2.29] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants at Each Score on the COVID Clinical Progression Scale at Day 14
Description: as for outcome 6
Time Frame: Day 14
Population: Participants with data collected at day 14.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 594 | 596
Participants
  0 = No clinical or virological evidence of infection | 21 | 28
  1 = No limitation of activities | 566 | 557
  2 = Limitation of activities | 7 | 11
  3 = Hospitalized, no oxygen therapy | 0 | 0
  4 = Hospitalized, on oxygen by mask or nasal prongs | 0 | 0
  5 = Hospitalized, on non-invasive ventilation or high-flow oxygen | 0 | 0
  6 = Hospitalized, on intubation and mechanical ventilation | 0 | 0
  7 = Hospitalized, on ventilation + additional organ support | 0 | 0
  8 = Death | 0 | 0
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; No hypothesis test or decision rule was evaluated; Test type: Superiority — Posterior probability of efficacy (P(OR<1)); Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.16 to 1.49] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants at Each Score on the COVID Clinical Progression Scale at Day 28
Description: as for outcome 6
Time Frame: Day 28
Population: Participants with data collected at day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 585 | 584
Participants
  0 = No clinical or virological evidence of infection | 17 | 22
  1 = No limitation of activities | 556 | 552
  2 = Limitation of activities | 11 | 10
  3 = Hospitalized, no oxygen therapy | 0 | 0
  4 = Hospitalized, on oxygen by mask or nasal prongs | 1 | 0
  5 = Hospitalized, on non-invasive ventilation or high-flow oxygen | 0 | 0
  6 = Hospitalized, on intubation and mechanical ventilation | 0 | 0
  7 = Hospitalized, on ventilation + additional organ support | 0 | 0
  8 = Death | 0 | 0
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; No hypothesis test or decision rule was evaluated; Test type: Superiority — Posterior probability of efficacy (P(OR<1)); Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.33 to 2.96] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Physical Function
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20, where a higher score correlates to better outcome for physical function.
Time Frame: Day 7, 14, 28, 90, 120, and 180
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
score on a scale
  Day 7: number analyzed (Participants) | 580 | 569
  Day 7 | 20 [19 to 20] | 20 [19 to 20]
  Day 14: number analyzed (Participants) | 570 | 564
  Day 14 | 20 [20 to 20] | 20 [20 to 20]
  Day 28: number analyzed (Participants) | 564 | 563
  Day 28 | 20 [20 to 20] | 20 [20 to 20]
  Day 90: number analyzed (Participants) | 552 | 544
  Day 90 | 20 [20 to 20] | 20 [20 to 20]
  Day 120: number analyzed (Participants) | 546 | 546
  Day 120 | 20 [20 to 20] | 20 [20 to 20]
  Day 180: number analyzed (Participants) | 415 | 414
  Day 180 | 20 [20 to 20] | 20 [20 to 20]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.71 to 1.31] — Initially estimated on the log relative odds scale, and then transformed to the odds ratio scale. On the log relative odds scale, the estimated parameter value was the posterior mean. Interval estimate is highest density Bayesian credible interval
Statistical Analysis 2: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.75 to 1.51] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.84 to 1.88] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.65 to 1.60] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 120; Test type: Other; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.57 to 1.36] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 180; Test type: Other; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.69 to 2.00] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Fatigue
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20, where a lower score correlates to better outcome for fatigue.
Time Frame: Day 7, 14, 28, 90, 120, and 180
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
score on a scale
  Day 7: number analyzed (Participants) | 580 | 571
  Day 7 | 4 [4 to 8] | 4 [4 to 8]
  Day 14: number analyzed (Participants) | 570 | 564
  Day 14 | 4 [4 to 7] | 4 [4 to 7]
  Day 28: number analyzed (Participants) | 565 | 563
  Day 28 | 4 [4 to 4] | 4 [4 to 5]
  Day 90: number analyzed (Participants) | 552 | 545
  Day 90 | 4 [4 to 4] | 4 [4 to 4]
  Day 120: number analyzed (Participants) | 546 | 547
  Day 120 | 4 [4 to 4] | 4 [4 to 4]
  Day 180: number analyzed (Participants) | 415 | 414
  Day 180 | 4 [4 to 4] | 4 [4 to 4]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.66 to 1.15] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.63 to 1.14] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.56 to 1.08] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.73 to 1.45] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 120; Test type: Other; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.71 to 1.40] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 180; Test type: Other; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.60 to 1.35] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Pain
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20, where a lower score correlates to better outcome for pain.
Time Frame: Day 7, 14, 28, 90, 120, and 180
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
score on a scale
  Day 7: number analyzed (Participants) | 579 | 570
  Day 7 | 4 [4 to 7] | 4 [4 to 7]
  Day 14: number analyzed (Participants) | 570 | 564
  Day 14 | 4 [4 to 4] | 4 [4 to 4]
  Day 28: number analyzed (Participants) | 564 | 563
  Day 28 | 4 [4 to 4] | 4 [4 to 4]
  Day 90: number analyzed (Participants) | 552 | 544
  Day 90 | 4 [4 to 4] | 4 [4 to 4]
  Day 120: number analyzed (Participants) | 546 | 547
  Day 120 | 4 [4 to 4] | 4 [4 to 4]
  Day 180: number analyzed (Participants) | 415 | 414
  Day 180 | 4 [4 to 4] | 4 [4 to 4]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.70 to 1.31] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.72 to 1.40] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.55 to 1.20] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.62 to 1.39] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 120; Test type: Other; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.65 to 1.46] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 180; Test type: Other; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.48 to 1.35] — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Depression
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domain with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20, where a lower score correlates to better outcome for depression.
Time Frame: Day 7, 14, 28, 90, 120, and 180
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
score on a scale
  Day 7: number analyzed (Participants) | 579 | 571
  Day 7 | 4 [4 to 4] | 4 [4 to 4]
  Day 14: number analyzed (Participants) | 570 | 564
  Day 14 | 4 [4 to 4] | 4 [4 to 4]
  Day 28: number analyzed (Participants) | 565 | 562
  Day 28 | 4 [4 to 4] | 4 [4 to 4]
  Day 90: number analyzed (Participants) | 552 | 545
  Day 90 | 4 [4 to 4] | 4 [4 to 4]
  Day 120: number analyzed (Participants) | 547 | 547
  Day 120 | 4 [4 to 4] | 4 [4 to 4]
  Day 180: number analyzed (Participants) | 415 | 413
  Day 180 | 4 [4 to 4] | 4 [4 to 4]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.62 to 1.24] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.65 to 1.38] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.49 to 1.13] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.67 to 1.55] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 120; Test type: Other; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.51 to 1.19] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 180; Test type: Other; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.49 to 1.35] — [estimate comment as in outcome 9, analysis 1]

13. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Anxiety
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20 where a lower score correlates to better outcome for anxiety.
Time Frame: Day 7, 14, 28, 90, 120, and 180
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
score on a scale
  Day 7: number analyzed (Participants) | 580 | 571
  Day 7 | 4 [4 to 5] | 4 [4 to 5]
  Day 14: number analyzed (Participants) | 570 | 564
  Day 14 | 4 [4 to 4] | 4 [4 to 4]
  Day 28: number analyzed (Participants) | 565 | 563
  Day 28 | 4 [4 to 4] | 4 [4 to 4]
  Day 90: number analyzed (Participants) | 552 | 544
  Day 90 | 4 [4 to 4] | 4 [4 to 4]
  Day 120: number analyzed (Participants) | 547 | 547
  Day 120 | 4 [4 to 4] | 4 [4 to 4]
  Day 180: number analyzed (Participants) | 415 | 414
  Day 180 | 4 [4 to 4] | 4 [4 to 4]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.77 to 1.41] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.82 to 1.69] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.52 to 1.14] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.65 to 1.43] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 120; Test type: Other; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.63 to 1.41] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 180; Test type: Other; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.44 to 1.19] — [estimate comment as in outcome 9, analysis 1]

14. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Social
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20 where a higher score correlates to better outcome for social roles and activities.
Time Frame: Day 7, 14, 28, 90, 120, and 180
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
score on a scale
  Day 7: number analyzed (Participants) | 580 | 569
  Day 7 | 20 [17 to 20] | 20 [16 to 20]
  Day 14: number analyzed (Participants) | 570 | 564
  Day 14 | 20 [20 to 20] | 20 [20 to 20]
  Day 28: number analyzed (Participants) | 564 | 563
  Day 28 | 20 [20 to 20] | 20 [20 to 20]
  Day 90: number analyzed (Participants) | 552 | 544
  Day 90 | 20 [20 to 20] | 20 [20 to 20]
  Day 120: number analyzed (Participants) | 547 | 547
  Day 120 | 20 [20 to 20] | 20 [20 to 20]
  Day 180: number analyzed (Participants) | 415 | 414
  Day 180 | 20 [20 to 20] | 20 [20 to 20]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.75 to 1.39] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.76 to 1.44] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.84 to 1.71] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.76 to 1.71] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 120; Test type: Other; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.67 to 1.46] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 180; Test type: Other; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.62 to 1.59] — [estimate comment as in outcome 9, analysis 1]

15. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Sleep
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20 where a lower score correlates to better outcome for sleep.
Time Frame: Day 7, 14, 28, 90, and 120
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 628 | 622
score on a scale
  Day 7: number analyzed (Participants) | 579 | 570
  Day 7 | 9 [8 to 10] | 9 [8 to 10]
  Day 14: number analyzed (Participants) | 570 | 564
  Day 14 | 9 [7 to 9] | 9 [7 to 9]
  Day 28: number analyzed (Participants) | 565 | 562
  Day 28 | 9 [7 to 9] | 9 [7 to 9]
  Day 90: number analyzed (Participants) | 552 | 543
  Day 90 | 8 [6 to 9] | 8 [6 to 9]
  Day 120: number analyzed (Participants) | 547 | 547
  Day 120 | 8 [6 to 9] | 8 [6 to 9]
  Day 180: number analyzed (Participants) | 415 | 414
  Day 180 | 8 [7 to 8] | 8 [6 to 9]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.74 to 1.14] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.79 to 1.22] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.71 to 1.08] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.80 to 1.21] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 120; Test type: Other; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.84 to 1.29] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Arm F - Montelukast vs Arm F - Placebo; Day 180; Test type: Other; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.68 to 1.14] — [estimate comment as in outcome 9, analysis 1]

16. Secondary Outcome: Time Unwell in Days as Measured by the Symptom and Clinical Event Scale
Description: The symptom and clinical event scale is a daily measurement that combines the global symptom burden scale with clinical events hospitalization and mortality. (No symptoms, mild symptoms, moderate symptoms, severe symptoms, hospitalized, deceased). Time unwell was the portion of follow-up (in days) that a participant was symptomatic, hospitalized, or deceased. The quantity is estimated from a Bayesian longitudinal ordinal regression model with covariate adjustment and weakly informative priors.
Time Frame: Up to 14 days
Population: Participants with data collected.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 618 | 610
days | 11.77 [11.58 to 11.97] | 12.01 [11.83 to 12.17]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; No hypothesis test or decision rule was evaluated; Test type: Superiority — Posterior probability of efficacy (P(Difference in MTU (Active - Placebo)<0)); Difference in model estimate time unwell = -0.24, 95% CI 2-sided [-0.6 to 0.1] — The mean time unwell is estimated from receipt of study drug to study day 14. The interval is a highest density credible interval

17. Secondary Outcome: Mean Days Benefit as Measured by the Symptom and Clinical Event Scale
Description: The symptom and clinical event scale is a daily measurement that combines the global symptom burden scale with clinical events hospitalization and mortality. (No symptoms, mild symptoms, moderate symptoms, severe symptoms, hospitalized, deceased). The cumulative benefit of treatment A is the probability of experiencing a better outcome on treatment A compared to treatment B, summed over the days of follow-up. The difference between the cumulative benefit of treatment A and the cumulative benefit of treatment B is known as the difference in days benefit. Measure of dispersion is 95% credible interval.
Time Frame: Up to 14 days
Population: Participants with data collected.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Arm F - Montelukast | Arm F - Placebo
Number analyzed (Participants) | 618 | 610
days | 3.25 [3.02 to 3.50] | 2.95 [2.72 to 3.16]
Statistical Analysis 1: Comparison: Arm F - Montelukast vs Arm F - Placebo; Analysis is exploratory. No hypothesis test or decision rule was evaluated; Test type: Superiority — Posterior probability of efficacy (P(Difference days benefit (Active - Placebo)>0)); Difference in model estimated means = 0.31, 95% CI 2-sided [-0.13 to 0.75] — The interval is a highest density credible interval

ADVERSE EVENTS:
Time Frame: Up to 180 days
Description: Participants were asked to complete daily assessments and report adverse events via the study portal through day 14, then at other intervals through day 28, and at follow up visits on day 90, 120, 180.
Arm/Group | Arm F - Montelukast | Arm F - Placebo
All-Cause Mortality (participants affected / at risk) | 0/628 | 0/622
Serious Adverse Events (participants affected / at risk) | 6/628 | 3/622
Other Adverse Events (participants affected / at risk) | 0/628 | 0/622
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm F - Montelukast (N=628) | Arm F - Placebo (N=622)
Pneumonia (Infections and infestations) | 1 | 1
Acute appendicitis (Gastrointestinal disorders) | 0 | 1
Cellulitis of legs (Skin and subcutaneous tissue disorders) | 1 | 0
Torsion of ovary (Reproductive system and breast disorders) | 1 | 0
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 | 0
Degloving injury (Skin and subcutaneous tissue disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture of calcaneus, open (Injury, poisoning and procedural complications) | 1 | 0
Paresthesia upper limb (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The first 202 participants to enroll to the montelukast study arm enrolled under protocol version 6, which only included follow-up through 120 days. The remainder of those enrolled to this study arm were consented to participate in the study up to 180 days. Of the 202 participants who enrolled under protocol version 6, two participants responded to Day 180 survey questions. Those participants are included in the Day 180 analysis to utilize all available responses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT05894577/Prot_001.pdf
  • Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT05894577/SAP_002.pdf
  • Informed Consent Form (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT05894577/ICF_000.pdf